CLINICAL TRIAL: NCT04457297
Title: A Randomized, Double-Blind, Phase III Study Comparing FTD/TPI Therapy Versus Placebo in Patients Who Are Positive for Blood Circulating Tumor DNA After Curative Resection of Colorectal Cancer
Brief Title: Initial Attack on Latent Metastasis Using TAS-102 for ct DNA Identified Colorectal Cancer Patients After Curative Resection
Acronym: ALTAIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Alpha-A, Inc. (Unknown)
Responsible Party: Principal Investigator, Takayuki Yoshino, MD., PhD Head of Department of Gastroenterology and Gastrointestinal Oncology, National Cancer Center Hospital East
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPOC 1905; JapicCTI-205363 (Registry Identifier: Japic Clinical Trials Information)
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Trifluridine and Tipiracil; Circulating Tumor DNA
Keywords: Colorectal Neoplasms; Gastrointestinal Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Antineoplastic Agents; trifluridine and tipiracil
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms; Digestive System Diseases; Gastrointestinal Diseases | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- trifluridine and tipiracil (Experimental)
  Interventions: Drug: trifluridine and tipiracil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: trifluridine and tipiracil — Trifluridine and tipiracil will be orally administered twice daily on Days 1 to 5 and Days 8 to 12. The administration will be repeated until completion of 6 courses(one course consists of 28 days) or until any discontinuation criterion is met.
  Arms: trifluridine and tipiracil
Drug: Placebo — Placebo will be orally administered twice daily on Days 1 to 5 and Days 8 to 12. The administration will be repeated until completion of 6 courses(one course consists of 28 days) or until any discontinuation criterion is met.
  Arms: Placebo

SUMMARY:
This trial is a randomized, double-blind, multinational Phase III study to evaluate the efficacy and safety of preemptive treatment with FTD/TPI compared with administration of placebo as follow-up, which is the standard of care, in patients who underwent curative resection of colorectal cancer and then tested positive for ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been histopathologically diagnosed with colorectal adenocarcinoma
2. Patients who have undergone radical curative resection of the primary and metastatic tumors
3. Patients with colon or rectal cancer of Stage III based on final findings (T any N1/2 M0) (UICC TNM Classification, 8th Edition) who have a past history of standard postoperative chemotherapy
4. Patients who tested positive for ctDNA using SignateraTM by an analysis of the latest blood samples collected within 3 months prior to enrollment
5. Patients with no obvious relapse confirmed by chest, abdominal, and pelvic CT scans, etc.
6. Patients who are capable of oral ingestion
7. Patients aged 20 years or older at the time of informed consent
8. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
9. Patients who have no severe disorder in major organs (such as the bone marrow, heart, lungs, liver, and kidneys) and meet the following criteria (Data obtained most recently and within 14 days of the date of enrollment will be used for enrollment. Data obtained 2 weeks before the date of enrollment, on the same day of the week as the enrollment date, may be used for enrollment.)

   * Neutrophil count ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * Hemoglobin ≥ 8.0 g/dL
   * Serum creatinine ≤ 1.5 mg/dL
   * Total bilirubin ≤ 1.5 mg/dL
   * ALT and AST ≤ 100 U/L
10. Patients with no diarrhea or stomatitis of Grade 2 or severer according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
11. Patients who voluntarily gave written consent to participate in the trial after receiving a thorough explanation of the trial before enrolling in the trial

Exclusion Criteria:

1. Patients with a history of treatment with FTD/TPI
2. Patients with a history of treatment with 2 or more regimens of postoperative adjuvant chemotherapy (Preoperative chemotherapy will not be counted as a regimen.)
3. Patients with a past history of a malignant tumor
4. Patients with a local or systemic active infection requiring intervention
5. Patients who are positive for HBs antigen or positive for HCV antibody
6. Patients who are positive for HIV antibody (Patients who have not been tested for HIV antibody may be enrolled.)
7. Patients with poorly controlled infections or diabetes
8. Patients with a past history of interstitial lung diseases (such as interstitial pneumonia and pulmonary fibrosis) requiring treatment or extensive findings of these diseases on CT
9. Patients with a serious complication
10. Patients who have been receiving systemic administration (oral or intravenous) of steroids (for 2 weeks or more at a dose of the equivalent of ≥ 10 mg/day of prednisolone)
11. Patients for whom enrollment in the trial is difficult because of clinically problematic psychiatric disorders
12. Pregnant or lactating women
13. Patients with reproductive potential who do not wish to use adequate contraceptive measures during the period of participation in the trial and during the contraception period
14. Patients who are judged by the attending physician to be ineligible for enrollment in the trial for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- Japan (38):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - University of Fukui Hospital, Yoshida, Fukui
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sano Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Kita, Kagawa-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - University Hospital, Kyoto Prefectural Univercity of Medicine, Kyoto, Kyoto
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Aizawa Hospital, Matsumoto, Nagano
  - Okayama University Hospital, Okayama, Okayama-ken
  - University of the Ryukyus Hospital, Nakagami, Okinawa
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saitama Cancer Center, Saitama, Saitama
  - Shimane Prefectural Central Hospital, Izumo, Shimane
  - Shizuoka Cancer Center, Shizuoka, Shizuoka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyo, Tokyo
  - National Cancer Center Hospital, Chūō, Tokyo
  - Cancer Institute Hospital Of JFCR, Koto, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Toyama University Hospital, Toyama, Toyama
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trifluridine and Tipiracil | Placebo
Started | 122 | 121
Completed | 122 | 121
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trifluridine and Tipiracil | Placebo | Total
Number analyzed (Participants) | 122 | 121 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 57 | 109
  >=65 years | 70 | 64 | 134
Age, Continuous [Median (Full Range); unit: years] | 67.0 [35 to 84] | 65.0 [34 to 86] | 66.0 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 71 | 70 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 122 | 121 | 243
Region of Enrollment [Number; unit: participants]
  Japan | 121 | 121 | 242
  Taiwan | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival 1 (DFS1)
Description: The time from the date of enrollment to any of the following events, whichever occurs first: a relapse, the first development of a secondary colorectal cancer lesion other than a relapse and death from any cause.
Time Frame: Up to 3 years
Population: Disease free survival 1 (DFS1) was assessed in Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
Months | 9.30 [7.82 to 10.84] | 5.55 [4.17 to 6.47]

2. Secondary Outcome: Rate of Conversion to Negative ctDNA
Description: This rate is defined as the proportion of subjects who became negative for ctDNA at the test immediately after completion of study treatment.
Time Frame: Up to 2 years
Population: Rate of Conversion to Negative ctDNA was assessed in Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
Percentage | 17.2 [11.0 to 25.1] | 12.4 [7.1 to 19.6]

3. Secondary Outcome: Disease-free Survival 2 (DFS2)
Description: The time from the date of enrollment to any of the following events, whichever occurs first: a relapse, development of a cancer lesion other than a relapse (secondary cancer), and death from any cause. For survives with no evidence of recurrence, DFS2 data will be censored at the last imaging date of confirmed no recurrence. Subjects for which no imaging have been performed, DFS2 data will be censored at the date of enrollment.
Time Frame: Up to 3 years
Population: Disease free survival 2 (DFS2) was assessed in Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
Months | 9.30 [7.82 to 10.84] | 5.55 [4.17 to 6.47]

4. Secondary Outcome: Overall Survival (OS)
Description: The time from the date of enrollment to the date of death from any cause. In surviving subjects, the last date of confirmation of survival will be treated as the end of this period. In subjects lost to follow-up, the last date of confirmation of survival before loss to follow-up will be treated as the end of this period.
Time Frame: Up to 3 years
Population: Overall survival (OS) was assessed in Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
Months | NA [NA to NA] — In the trifluridine and tipiracil group, because the number of events did not reach 50%, the median OS (95% CI) was not reach. | 37.26 [NA to NA] — In the placebo group, an event occurred in the patient with the longest follow-up period, allowing the median to be calculated. However, due to an insufficient number of events, the upper and lower limits of the confidence interval could not be calculated.

5. Secondary Outcome: Treatment Completion Rate
Description: This rate had calculated for each eligible subject in accordance with the following equation: Treatment completion rate (%) = number of treatment courses completed/6 × 100
Time Frame: Up to 3 years
Population: Treatment completion rate was assessed in Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Percentage of treatment completion
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
Percentage of treatment completion | 77.87 (30.26) | 78.79 (25.46)

6. Secondary Outcome: QOL (Week 24 Only)
Description: Measure Description:
  Quality of Life was assessed using two validated instruments:
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) evaluates cancer-specific HRQoL across domains:
  Global Health Status/QoL (range: 0-100, higher = better global health/QoL), Functional Scales (Physical, Role, Emotional, Cognitive, Social; each range: 0-100, higher = better functioning), Symptom Scales (Fatigue, Nausea/vomiting, Pain, Dyspnoea, Insomnia, Appetite loss, Constipation, Diarrhoea, Financial difficulties): each 0-100 (higher = worse/more severe symptoms).
  Scores are linearly transformed; subscales are reported individually (not summed).
  EQ-5D-5L (EuroQOL 5-Dimension 5-Level) measures general health across five dimensions:
  Index Score (range: -1.000 to 1.000, higher = better health), Visual Analogue Scale (VAS) (range: 0-100, higher = better health). Unit of Measure: scores on a scale. Note: Only Week 24 results are presented.
Time Frame: Up to 1 year
Population: QOL was assessed in Full Analysis Set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Trifluridine and Tipiracil | Placebo
Number analyzed (Participants) | 122 | 121
scores on a scale
  Global healthstatus/QoL (Week 24) | 0.00 (22.71) | 4.36 (22.39)
  EORTC QLQ-C30 Functional scales: Physical functioning (Week 24) | -1.10 (13.64) | 1.13 (9.47)
  EORTC QLQ-C30 Functional scales: Role functioning (Week 24) | -3.33 (14.27) | -3.33 (12.57)
  EORTC QLQ-C30 Functional scales: Emotional functioning (Week 24) | 4.22 (14.86) | 0.64 (13.84)
  EORTC QLQ-C30 Functional scales: Cognitive functioning (Week 24) | 0.20 (15.75) | 2.56 (17.49)
  EORTC QLQ-C30 Functional scales: Social functioning (Week 24) | -2.55 (12.99) | 1.28 (12.95)
  EORTC QLQ-C30 Symptom scales: Fatigue (Week 24) | 3.14 (16.76) | -2.74 (16.90)
  EORTC QLQ-C30 Symptom scales: Nausea and vomiting (Week 24) | 4.12 (1.28) | 10.26 (7.96)
  EORTC QLQ-C30 Symptom scales: Pain (Week 24) | -1.18 (15.17) | 1.54 (15.23)
  EORTC QLQ-C30 Symptom scales: Dyspnoea (Week 24) | 1.18 (18.86) | 0.51 (17.17)
  EORTC QLQ-C30 Symptom scales: Insomnia (Week 24) | -0.39 (25.46) | -0.51 (15.01)
  EORTC QLQ-C30 Symptom scales: Appetite (Week 24) | 5.49 (21.73) | 1.03 (13.14)
  EORTC QLQ-C30 Symptom scales: Constipation (Week 24) | 2.75 (20.71) | 3.08 (20.18)
  EORTC QLQ-C30 Symptom scales: Diarrhoea (Week 24) | 6.67 (22.30) | 4.62 (22.15)
  EORTC QLQ-C30 Symptom scales: Financial difficulties (Week 24) | -4.31 (21.07) | -2.05 (20.31)
  EQ-5D-5L Index Score (Week 24) | -0.0019 (0.0170) | 0.1110 (0.0986)
  EQ-5D-5L VAS (Week 24) | 1.2 (12.7) | 1.6 (13.0)

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Trifluridine and Tipiracil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/121
Serious Adverse Events (participants affected / at risk) | 6/122 | 0/121
Other Adverse Events (participants affected / at risk) | 120/122 | 69/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trifluridine and Tipiracil (N=122) | Placebo (N=121)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trifluridine and Tipiracil (N=122) | Placebo (N=121)
Anaemia (Blood and lymphatic system disorders) | 32 | 2
Neutropenia (Blood and lymphatic system disorders) | 15 | 0
Decreased appetite (Metabolism and nutrition disorders) | 27 | 2
Dysgeusia (Nervous system disorders) | 10 | 1
Headache (Nervous system disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 41 | 13
Nausea (Gastrointestinal disorders) | 63 | 15
Stomatitis (Gastrointestinal disorders) | 18 | 7
Vomiting (Gastrointestinal disorders) | 12 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 0
Fatigue (General disorders) | 18 | 6
Malaise (General disorders) | 19 | 7
Pyrexia (General disorders) | 8 | 4
Blood bilirubin increased (Investigations) | 9 | 5
Lymphocyte count decreased (Investigations) | 10 | 1
Neutrophil count decreased (Investigations) | 91 | 5
Platelet count decreased (Investigations) | 15 | 4
White blood cell count decreased (Investigations) | 78 | 4
Leukopenia (Blood and lymphatic system disorders) | 8 | 0
Constipation (Gastrointestinal disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT04457297/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT04457297/SAP_001.pdf